CLINICAL TRIAL: NCT02464930
Title: Evaluation of MicroRNA Expression in Blood and Cytology Specimens as a Novel Method for Detecting Barrett's Esophagus
Brief Title: Evaluation of MicroRNA Expression in Blood and Cytology for Detecting Barrett's Esophagus and Associated Neoplasia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Midwest Biomedical Research Foundation (Other)
Collaborators: Kansas City Veteran Affairs Medical Center (U.S. Federal Agency); University of Kansas (Other)
Responsible Party: Principal Investigator, Ajay Bansal, Associate Professor of Medicine and Staff Gastroenterologist, Midwest Biomedical Research Foundation
Organization: Midwest Veterans' Biomedical Research Foundation (Other)
Other Study IDs: AB0009
Record Dates: First submitted 2015-06-02; First posted 2015-06-08 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Barrett's Esophagus; Gastroesophageal Reflux; Esophageal Adenocarcinoma
Keywords: Blood; Cytology; Esophagus; microRNA
MeSH Terms: conditions — Barrett Esophagus; Gastroesophageal Reflux; Adenocarcinoma Of Esophagus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, bile and tissue in a repository
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- No-GERD Controls: NERD controls will be enrolled from subjects presenting to the endoscopy unit who are being evaluated for reasons other than GERD or BE surveillance. These are patients who are referred to the endoscopy unit for: evaluation of anemia, dysphagia, occult blood positivity, gastrointestinal blood loss etc.
  * No history of GERD
  * Response "no" to presence of symptoms on a standardized GERD questionnaire
  * No prescriptions for acid suppressive medication over the past 2 years as documented in electronic pharmacy records.
  * Normal endoscopy that does not find Barrett's esophagus, hiatus hernia or erosive esophagitis.
- GERD Controls: * Respond "yes" to the presence of symptoms on a standardized GERD questionnaire
  * Prescriptions for acid suppressive medication as documented in electronic pharmacy records.
- BE Cases: • Patients who present for evaluation of reflux symptoms and are found to have at least 1 cm of columnar lined esophagus on endoscopy with intestinal metaplasia on biopsies. This will include patients with esophageal adenocarcinoma

SUMMARY:
The primary purpose of this study is to test new methods to diagnose BE in time before it turns into advanced cancer. Once BE is diagnosed, the current standard of care is to monitor the disease so that complication such as cancer can be diagnosed early. The two new methods the investigators are evaluating are: a) blood test and b) brush test of the food pipe. The investigators will collect blood, bile and cells from the food pipe and stomach and measure for a biomarker called microRNA (miRNA). In the future, measurements of microRNA biomarkers could help the doctors figure out which patients are at increased risk for cancer of the esophagus.

DETAILED DESCRIPTION:
The investigators will collect serum, bile and esophageal cells (using cytology devices) from consenting subjects. The investigators have previously identified BE specific miRNA that will be tested on the cytology specimens. These are miRNAs -192-5p, -215-5p and -194-5p. The investigators have also identified serum microRNAs in whole serum and exosomes by sequencing to study further. The investigators will also evaluate miRNA expression within biliary exosomes for the first time in patients with reflux related diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patient age: > 18 years
* Ability to provide written, informed consent

Exclusion Criteria:

* Pregnancy or planning a pregnancy
* History of nasal, esophageal & gastric surgery
* History of recurrent epistaxis or nasal trauma
* Subjects with a history of unresolved drug or alcohol dependency
* Inability to obtain biopsies due to a coagulopathy, varices, thrombocytopenia, etc.
* Subjects with inadequate cytology specimens will not undergo repeat test and will be excluded from the study
* Inability to provide written informed consent
* Inability to discontinue drugs such as Plavix
* Advanced chronic liver disease
* Severe uncontrolled coagulopathy
* Active cancer in any organ over the past 3 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited at the Kansas City VA Hospital and the Mobile Medical unit of the Kansas City VA. The Mobile Medical Unit (MMU) travels to multiple counties to provide health care to the veterans at their doorstep. This is a program that has been in place for several years and continues to grow. Currently, the MMU provides services such as basic health evaluations and phlebotomy to ~600 veterans per week.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2015-04; Primary Completion 2018-04 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of tissue and serum microRNA expression by digital polymerase chain reaction for diagnosis of BE neoplasia | 1-3 years
  The two main outcomes are the diagnostic accuracy of tissue and serum microRNA for the the diagnosis of Barrett's esophagus compared to endoscopy.

SECONDARY OUTCOMES:
Differences in the microRNA expression of biliary exosomes between GERD, Barrett's esophagus and Cancer | 1-3 years
  The microRNA expression will be measured by digital polymerase chain reaction

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Bansal, MD, Principal Investigator — Veterans Affairs Medical Center and the University of Kansas Medical Center
Locations (1):
- Kansas City Veterans Affairs Medical Center, Kansas City, Missouri, United States

REFERENCES:
- [Background] El-Serag HB, Sweet S, Winchester CC, Dent J. Update on the epidemiology of gastro-oesophageal reflux disease: a systematic review. Gut. 2014 Jun;63(6):871-80. doi: 10.1136/gutjnl-2012-304269. Epub 2013 Jul 13. PMID 23853213
- [Background] Spechler SJ, Souza RF. Barrett's esophagus. N Engl J Med. 2014 Aug 28;371(9):836-45. doi: 10.1056/NEJMra1314704. No abstract available. PMID 25162890
- [Background] Rajendra S, Sharma P. Barrett's Esophagus. Curr Treat Options Gastroenterol. 2014 Jun;12(2):169-82. doi: 10.1007/s11938-014-0012-0. PMID 24634008
- [Background] Weaver JMJ, Ross-Innes CS, Shannon N, Lynch AG, Forshew T, Barbera M, Murtaza M, Ong CJ, Lao-Sirieix P, Dunning MJ, Smith L, Smith ML, Anderson CL, Carvalho B, O'Donovan M, Underwood TJ, May AP, Grehan N, Hardwick R, Davies J, Oloumi A, Aparicio S, Caldas C, Eldridge MD, Edwards PAW, Rosenfeld N, Tavare S, Fitzgerald RC; OCCAMS consortium. Ordering of mutations in preinvasive disease stages of esophageal carcinogenesis. Nat Genet. 2014 Aug;46(8):837-843. doi: 10.1038/ng.3013. Epub 2014 Jun 22. PMID 24952744
- [Background] Hamilton SR, Smith RR, Cameron JL. Prevalence and characteristics of Barrett esophagus in patients with adenocarcinoma of the esophagus or esophagogastric junction. Hum Pathol. 1988 Aug;19(8):942-8. doi: 10.1016/s0046-8177(88)80010-8. PMID 3402983
- [Background] di Pietro M, Alzoubaidi D, Fitzgerald RC. Barrett's esophagus and cancer risk: how research advances can impact clinical practice. Gut Liver. 2014 Jul;8(4):356-70. doi: 10.5009/gnl.2014.8.4.356. Epub 2014 Jul 1. PMID 25071900
- [Background] American Gastroenterological Association; Spechler SJ, Sharma P, Souza RF, Inadomi JM, Shaheen NJ. American Gastroenterological Association medical position statement on the management of Barrett's esophagus. Gastroenterology. 2011 Mar;140(3):1084-91. doi: 10.1053/j.gastro.2011.01.030. No abstract available. PMID 21376940
- [Background] Sharma P. Clinical practice. Barrett's esophagus. N Engl J Med. 2009 Dec 24;361(26):2548-56. doi: 10.1056/NEJMcp0902173. No abstract available. PMID 20032324
- [Background] Hur C, Miller M, Kong CY, Dowling EC, Nattinger KJ, Dunn M, Feuer EJ. Trends in esophageal adenocarcinoma incidence and mortality. Cancer. 2013 Mar 15;119(6):1149-58. doi: 10.1002/cncr.27834. Epub 2012 Dec 11. PMID 23303625
- [Background] Yousef F, Cardwell C, Cantwell MM, Galway K, Johnston BT, Murray L. The incidence of esophageal cancer and high-grade dysplasia in Barrett's esophagus: a systematic review and meta-analysis. Am J Epidemiol. 2008 Aug 1;168(3):237-49. doi: 10.1093/aje/kwn121. Epub 2008 Jun 12. PMID 18550563
- [Background] Hvid-Jensen F, Pedersen L, Drewes AM, Sorensen HT, Funch-Jensen P. Incidence of adenocarcinoma among patients with Barrett's esophagus. N Engl J Med. 2011 Oct 13;365(15):1375-83. doi: 10.1056/NEJMoa1103042. PMID 21995385
- [Background] Reid BJ, Li X, Galipeau PC, Vaughan TL. Barrett's oesophagus and oesophageal adenocarcinoma: time for a new synthesis. Nat Rev Cancer. 2010 Feb;10(2):87-101. doi: 10.1038/nrc2773. PMID 20094044
- [Background] Montgomery E, Goldblum JR, Greenson JK, Haber MM, Lamps LW, Lauwers GY, Lazenby AJ, Lewin DN, Robert ME, Washington K, Zahurak ML, Hart J. Dysplasia as a predictive marker for invasive carcinoma in Barrett esophagus: a follow-up study based on 138 cases from a diagnostic variability study. Hum Pathol. 2001 Apr;32(4):379-88. doi: 10.1053/hupa.2001.23511. PMID 11331954
- [Background] Shaheen NJ, Hur C. Garlic, silver bullets, and surveillance upper endoscopy for Barrett's esophagus. Gastroenterology. 2013 Aug;145(2):273-6. doi: 10.1053/j.gastro.2013.06.028. Epub 2013 Jun 24. No abstract available. PMID 23806540
- [Background] Kadri SR, Lao-Sirieix P, O'Donovan M, Debiram I, Das M, Blazeby JM, Emery J, Boussioutas A, Morris H, Walter FM, Pharoah P, Hardwick RH, Fitzgerald RC. Acceptability and accuracy of a non-endoscopic screening test for Barrett's oesophagus in primary care: cohort study. BMJ. 2010 Sep 10;341:c4372. doi: 10.1136/bmj.c4372. PMID 20833740
- [Background] Bansal A, Lee IH, Hong X, Anand V, Mathur SC, Gaddam S, Rastogi A, Wani SB, Gupta N, Visvanathan M, Sharma P, Christenson LK. Feasibility of mcroRNAs as biomarkers for Barrett's Esophagus progression: a pilot cross-sectional, phase 2 biomarker study. Am J Gastroenterol. 2011 Jun;106(6):1055-63. doi: 10.1038/ajg.2011.37. Epub 2011 Mar 15. PMID 21407181
- [Background] Bhardwaj A, Hollenbeak CS, Pooran N, Mathew A. A meta-analysis of the diagnostic accuracy of esophageal capsule endoscopy for Barrett's esophagus in patients with gastroesophageal reflux disease. Am J Gastroenterol. 2009 Jun;104(6):1533-9. doi: 10.1038/ajg.2009.86. Epub 2009 Apr 21. PMID 19491867
- [Background] Gora MJ, Sauk JS, Carruth RW, Lu W, Carlton DT, Soomro A, Rosenberg M, Nishioka NS, Tearney GJ. Imaging the upper gastrointestinal tract in unsedated patients using tethered capsule endomicroscopy. Gastroenterology. 2013 Oct;145(4):723-5. doi: 10.1053/j.gastro.2013.07.053. Epub 2013 Aug 8. No abstract available. PMID 23932950
- [Background] Benaglia T, Sharples LD, Fitzgerald RC, Lyratzopoulos G. Health benefits and cost effectiveness of endoscopic and nonendoscopic cytosponge screening for Barrett's esophagus. Gastroenterology. 2013 Jan;144(1):62-73.e6. doi: 10.1053/j.gastro.2012.09.060. Epub 2012 Oct 3. PMID 23041329
- [Background] Rajewsky N. microRNA target predictions in animals. Nat Genet. 2006 Jun;38 Suppl:S8-13. doi: 10.1038/ng1798. PMID 16736023
- [Background] Cortez MA, Bueso-Ramos C, Ferdin J, Lopez-Berestein G, Sood AK, Calin GA. MicroRNAs in body fluids--the mix of hormones and biomarkers. Nat Rev Clin Oncol. 2011 Jun 7;8(8):467-77. doi: 10.1038/nrclinonc.2011.76. PMID 21647195
- [Background] Liu N, Chen NY, Cui RX, Li WF, Li Y, Wei RR, Zhang MY, Sun Y, Huang BJ, Chen M, He QM, Jiang N, Chen L, Cho WC, Yun JP, Zeng J, Liu LZ, Li L, Guo Y, Wang HY, Ma J. Prognostic value of a microRNA signature in nasopharyngeal carcinoma: a microRNA expression analysis. Lancet Oncol. 2012 Jun;13(6):633-41. doi: 10.1016/S1470-2045(12)70102-X. Epub 2012 May 3. PMID 22560814
- [Background] Lu J, Getz G, Miska EA, Alvarez-Saavedra E, Lamb J, Peck D, Sweet-Cordero A, Ebert BL, Mak RH, Ferrando AA, Downing JR, Jacks T, Horvitz HR, Golub TR. MicroRNA expression profiles classify human cancers. Nature. 2005 Jun 9;435(7043):834-8. doi: 10.1038/nature03702. PMID 15944708
- [Background] Wang S, Wang L, Bayaxi N, Li J, Verhaegh W, Janevski A, Varadan V, Ren Y, Merkle D, Meng X, Gao X, Wang H, Ren J, Kuo WP, Dimitrova N, Wu Y, Zhu H. A microRNA panel to discriminate carcinomas from high-grade intraepithelial neoplasms in colonoscopy biopsy tissue. Gut. 2013 Feb;62(2):280-9. doi: 10.1136/gutjnl-2011-301554. Epub 2012 Apr 25. PMID 22535378
- [Background] Lujambio A, Lowe SW. The microcosmos of cancer. Nature. 2012 Feb 15;482(7385):347-55. doi: 10.1038/nature10888. PMID 22337054
- [Background] Raposo G, Stoorvogel W. Extracellular vesicles: exosomes, microvesicles, and friends. J Cell Biol. 2013 Feb 18;200(4):373-83. doi: 10.1083/jcb.201211138. PMID 23420871
- [Background] Zaidi AH, Gopalakrishnan V, Kasi PM, Zeng X, Malhotra U, Balasubramanian J, Visweswaran S, Sun M, Flint MS, Davison JM, Hood BL, Conrads TP, Bergman JJ, Bigbee WL, Jobe BA. Evaluation of a 4-protein serum biomarker panel-biglycan, annexin-A6, myeloperoxidase, and protein S100-A9 (B-AMP)-for the detection of esophageal adenocarcinoma. Cancer. 2014 Dec 15;120(24):3902-13. doi: 10.1002/cncr.28963. Epub 2014 Aug 5. PMID 25100294
- [Background] Varghese S, Lao-Sirieix P, Fitzgerald RC. Identification and clinical implementation of biomarkers for Barrett's esophagus. Gastroenterology. 2012 Mar;142(3):435-441.e2. doi: 10.1053/j.gastro.2012.01.013. Epub 2012 Jan 20. No abstract available. PMID 22266150
- [Background] Garman KS, Owzar K, Hauser ER, Westfall K, Anderson BR, Souza RF, Diehl AM, Provenzale D, Shaheen NJ. MicroRNA expression differentiates squamous epithelium from Barrett's esophagus and esophageal cancer. Dig Dis Sci. 2013 Nov;58(11):3178-88. doi: 10.1007/s10620-013-2806-7. Epub 2013 Aug 8. PMID 23925817
- [Background] Sakai NS, Samia-Aly E, Barbera M, Fitzgerald RC. A review of the current understanding and clinical utility of miRNAs in esophageal cancer. Semin Cancer Biol. 2013 Dec;23(6 Pt B):512-21. doi: 10.1016/j.semcancer.2013.08.005. Epub 2013 Sep 3. PMID 24013023
- [Background] Talsma AK, Ong CA, Liu X, van Hagen P, Van Lanschot JJ, Tilanus HW, Hardwick RH, Carroll NR, Spaander MC, Fitzgerald RC, Wijnhoven BP. Location of lymph node involvement in patients with esophageal adenocarcinoma predicts survival. World J Surg. 2014 Jan;38(1):106-13. doi: 10.1007/s00268-013-2236-x. PMID 24101018
- [Background] Wang K, Zhang S, Marzolf B, Troisch P, Brightman A, Hu Z, Hood LE, Galas DJ. Circulating microRNAs, potential biomarkers for drug-induced liver injury. Proc Natl Acad Sci U S A. 2009 Mar 17;106(11):4402-7. doi: 10.1073/pnas.0813371106. Epub 2009 Feb 25. PMID 19246379
- [Background] Wang WS, Liu LX, Li GP, Chen Y, Li CY, Jin DY, Wang XL. Combined serum CA19-9 and miR-27a-3p in peripheral blood mononuclear cells to diagnose pancreatic cancer. Cancer Prev Res (Phila). 2013 Apr;6(4):331-8. doi: 10.1158/1940-6207.CAPR-12-0307. Epub 2013 Feb 19. PMID 23430754
- [Background] Weiland M, Gao XH, Zhou L, Mi QS. Small RNAs have a large impact: circulating microRNAs as biomarkers for human diseases. RNA Biol. 2012 Jun;9(6):850-9. doi: 10.4161/rna.20378. Epub 2012 Jun 1. PMID 22699556
- [Background] Arroyo JD, Chevillet JR, Kroh EM, Ruf IK, Pritchard CC, Gibson DF, Mitchell PS, Bennett CF, Pogosova-Agadjanyan EL, Stirewalt DL, Tait JF, Tewari M. Argonaute2 complexes carry a population of circulating microRNAs independent of vesicles in human plasma. Proc Natl Acad Sci U S A. 2011 Mar 22;108(12):5003-8. doi: 10.1073/pnas.1019055108. Epub 2011 Mar 7. PMID 21383194
- [Background] Beg MS, Navaneethan U, Atiq M, Komrokji R, Safa M. Outcome of esophageal carcinoma in the veteran affairs population: a comparative analysis from the Veteran Affairs Central Cancer Registry. Am J Clin Oncol. 2009 Jun;32(3):286-90. doi: 10.1097/COC.0b013e31818af0d8. PMID 19433959
- [Background] Lao-Sirieix P, Boussioutas A, Kadri SR, O'Donovan M, Debiram I, Das M, Harihar L, Fitzgerald RC. Non-endoscopic screening biomarkers for Barrett's oesophagus: from microarray analysis to the clinic. Gut. 2009 Nov;58(11):1451-9. doi: 10.1136/gut.2009.180281. Epub 2009 Aug 2. PMID 19651633
- [Background] Wang KK, Sampliner RE; Practice Parameters Committee of the American College of Gastroenterology. Updated guidelines 2008 for the diagnosis, surveillance and therapy of Barrett's esophagus. Am J Gastroenterol. 2008 Mar;103(3):788-97. doi: 10.1111/j.1572-0241.2008.01835.x. No abstract available. PMID 18341497
- [Background] Sharma P, Dent J, Armstrong D, Bergman JJ, Gossner L, Hoshihara Y, Jankowski JA, Junghard O, Lundell L, Tytgat GN, Vieth M. The development and validation of an endoscopic grading system for Barrett's esophagus: the Prague C & M criteria. Gastroenterology. 2006 Nov;131(5):1392-9. doi: 10.1053/j.gastro.2006.08.032. Epub 2006 Aug 16. PMID 17101315
- [Background] Tuck MK, Chan DW, Chia D, Godwin AK, Grizzle WE, Krueger KE, Rom W, Sanda M, Sorbara L, Stass S, Wang W, Brenner DE. Standard operating procedures for serum and plasma collection: early detection research network consensus statement standard operating procedure integration working group. J Proteome Res. 2009 Jan;8(1):113-7. doi: 10.1021/pr800545q. PMID 19072545
- [Background] Montgomery E, Bronner MP, Goldblum JR, Greenson JK, Haber MM, Hart J, Lamps LW, Lauwers GY, Lazenby AJ, Lewin DN, Robert ME, Toledano AY, Shyr Y, Washington K. Reproducibility of the diagnosis of dysplasia in Barrett esophagus: a reaffirmation. Hum Pathol. 2001 Apr;32(4):368-78. doi: 10.1053/hupa.2001.23510. PMID 11331953
- [Background] Bansal A, Lee IH, Hong X, Mathur SC, Tawfik O, Rastogi A, Buttar N, Visvanathan M, Sharma P, Christenson LK. Discovery and validation of Barrett's esophagus microRNA transcriptome by next generation sequencing. PLoS One. 2013;8(1):e54240. doi: 10.1371/journal.pone.0054240. Epub 2013 Jan 23. PMID 23372692
- [Background] Schisterman EF, Perkins NJ, Liu A, Bondell H. Optimal cut-point and its corresponding Youden Index to discriminate individuals using pooled blood samples. Epidemiology. 2005 Jan;16(1):73-81. doi: 10.1097/01.ede.0000147512.81966.ba. PMID 15613948